CLINICAL TRIAL: NCT00003041
Title: Phase II Evaluation of Pyrazoloacridine (NSC #366140) in Patients With Metastatic Breast Cancer
Brief Title: Pyrazoloacridine in Treating Women With Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065670; OSU-9712; NCI-T96-0120
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2002-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — NSC 366140

INTERVENTIONS:
Drug: pyrazoloacridine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of pyrazoloacridine in treating women who have refractory metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of pyrazoloacridine in patients with refractory breast cancer. II. Determine the toxic effects of pyrazoloacridine in these patients.

OUTLINE: Patients receive pyrazoloacridine IV over 3 hours. Treatment repeats every 21 days for 2-8 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic breast cancer Bidimensionally measurable disease of any of the following types required: Bidimensionally measurable lung lesions on chest X-ray, CT scan, or MRI Palpable and quantifiable lymph nodes at least 2 x 2 cm Abdominal mass at least 2 x 2 cm quantifiable by CT scan Bidimensionally measurable liver metastases at least 2 x 2 cm Palpable hepatomegaly if liver edge is clearly defined and extends at least 5 cm below the costal margin of the xiphoid process Unacceptable as measurable disease: Diffuse lung infiltration or unidimensionally measurable hilar lesions Pelvic mass of indefinite dimension Bone metastases Pleural effusion or ascites No brain metastases Must have failed or progressed on prior therapy or relapsed less than 12 months after therapy discontinuation Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 16 and over Sex: Female Menopausal status: Not specified Performance status: SWOG 0-2 Life expectancy: At least 6 months Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT no greater than 2.5 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of congestive heart failure, myocardial infarction within past 6 months, ventricular arrhythmia, or ischemic heart disease requiring medication If necessary, ejection fraction at least 50% by MUGA Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other prior malignancies in past 5 years other than basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix No other serious illnesses or active infections No seizure disorder requiring anticonvulsant therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: See Disease Characteristics No more than 2 prior chemotherapy regimens for metastatic disease One prior adjuvant chemotherapy regimen for metastatic disease allowed At least 4 weeks since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: One prior regimen of hormonal therapy for metastatic disease allowed At least 3 weeks since prior hormonal therapy and recovered No concurrent hormonal or corticosteroid therapy Radiotherapy: At least 4 weeks since prior radiotherapy to less than 25% bone marrow No concurrent radiotherapy Surgery: At least 4 weeks since prior surgery and recovered No concurrent surgery Other: At least 4 weeks since any prior treatment directed at the tumor and recovered No other concurrent anticancer or investigational therapy No concurrent participation on another therapeutic clinical trial

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric H. Kraut, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Central Baptist Hospital, Lexington, Kentucky
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Grant/Riverside Methodist Hospitals, Columbus, Ohio
  - Mount Carmel, Columbus, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina